CLINICAL TRIAL: NCT05984147
Title: A Phase 1, Open Label, Dose Escalation, Dose Expansion, Multicenter Study Evaluating the Safety, Pharmacokinetics and Pharmacodynamics of Oral AUR108 in Patients With Relapsed Advanced Lymphomas(ASHA-1)
Brief Title: A Study Evaluating the Safety and Efficacy of AUR108 in Patients With Relapsed Advanced Lymphomas (ASHA-1)
Acronym: ASHA-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aurigene Discovery Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AUR108-101
Record Dates: First submitted 2023-07-20; First posted 2023-08-09 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Relapsed Advanced Lymphomas
Keywords: Relapse Advanced Lymphomas; Diffuse large B-cell lymphoma; Follicular lymphoma; Mature T/NK-cell lymphomas; Other Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, T-Cell

STUDY DESIGN:
Intervention Model Description: Sequential Assignment Dose Escalation "3+3" Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AUR108, 50mg to 300mg (Experimental): Currently, planned dose levels are 50,90,150,220,300 mg will be administered in 3+/4- regimen.
  Interventions: Drug: AUR108

INTERVENTIONS:
Drug: AUR108 — 3 Days dosing, and 4 days no dose in a week

SUMMARY:
An open-label, first-in-human, Phase 1 study in adult patients with relapsed advanced lymphomas will be done to assess AUR108 safety, tolerability, pharmacokinetics, pharmacodynamics, and optimal biological dose.

DETAILED DESCRIPTION:
This is a Phase I, Open Label, Dose-Escalation, First-in-Human study in adult patients with select relapsed advanced lymphomas. The safety and tolerability of oral AUR108 will be evaluated in patients with Non-Hodgkin lymphoma and Hodgkin lymphoma who do not have any available curative or life-prolonging treatment options and have exhausted all effective locally available therapies. The traditional 3+3 design for dose escalation will be used to evaluate the safety, pharmacokinetics/pharmacodynamics, and determine the Optimal Biological Dose of AUR108 as a single agent. The Optimal Biological Dose will be selected using a totality of safety, PK, and PD data.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 years of age
2. Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1
3. Acceptable bone marrow and organ function at screening as described below:

   1. ANC ≥ 1000/μL (without WBC growth factor support)
   2. Platelet count ≥ 75,000/μL without transfusion support
   3. Hemoglobin ≥ 9 g/dL (Transfusion is allowed to achieve this Hb)
   4. Total Bilirubin ≤ 1.5 x ULN; (Patients with known Gilbert's syndrome are allowed with a Total Bilirubin ≤ 2.5 x ULN)
   5. AST (SGOT) ≤ 3 x ULN (≤ 5 × ULN if known liver metastases)
   6. ALT (SGPT) ≤ 3 x ULN (≤ 5 × ULN if known liver metastases)
   7. Creatinine clearance (CrCl) ≥ 30 mL/min (either measured or estimated by the Cockcroft-Gault formula). (Cockcroft-Gault formula for estimated creatinine clearance [eCrCl]: eCrCl = [140- Age] × Weight [kg] × [0.85 if Female] / [72 × serum creatinine (mg/dL)]).
4. Ability to swallow and retain oral medications
5. Histo-pathological diagnosis of a Non-Hodgkin lymphoma orHodgkin Lymphoma. Note: The lymphoma should be either in Stage III or IV according to Lugano classification (Cheson BD et al, 2014) at screening.
6. In the case of subjects who have lymphoma for which high-dose chemotherapy and autologous stem cell transplantation (HDASCT) is considered a standard curative therapy, eligibility for this study requires that the subject's disease has relapsed after HDASCT, that the subject is not eligible for HD-ASCT, or that the subject has refused HD-ASCT.
7. In the case of subjects who have lymphoma for which CAR-T therapy is considered a standard therapy, eligibility for this study requires that the subjects disease has relapsed after CAR-T, or that the subject has refused CAR-T, or that the CAR-T therapy is not accessible to the patient.
8. Evidence of measurable disease as per Lugano Criteria for Lymphoma (Cheson BD et al, 2014).
9. Standard curative measures do not exist, and patient must have exhausted all effective therapies, available locally.

   1. At a minimum, the patients must have received at least 2 prior lines of systemic therapies. These systemic therapies could be either in the stage II, III or IV.
   2. Any cancer patient with access to any effective therapy must not be enrolled.

Exclusion Criteria:

1. Systemic anti-cancer therapy, such as chemotherapy, or biological therapy, immunomodulatory drug therapy, received within the past 28 days or 5 half-lives, whichever is longer, from the Cycle 1 Day 1 of the study.

   Note: Concomitant use of low dose prednisone (up to 10 mg/day) is allowed.
2. Presence of an acute or chronic toxicity resulting from prior anticancer treatment, with the exception of alopecia or nail changes, that has not resolved to Grade ≤ 1, as determined by NCI CTCAE v 5.0.
3. Definitive Radiotherapy within the last 21 days of Cycle 1 Day 1 (limited field palliative radiation is allowed and no restrictions during the screening period or during the trial).
4. Use of any investigational agent within 28 days or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1.
5. Patients with cutaneous lymphomas, mycosis fungoides (MF) or Sézary syndrome (SS).
6. Primary CNS lymphoma
7. Known symptomatic or untreated or recently treated (≤ 6 months of screening) central nervous system (CNS) lymphoma. Patients with previously treated (> 6 months of screening) CNS lymphoma and are now stable and asymptomatic, from CNS perspective, are allowed
8. Patients with lymphoma that requires immediate cytoreductive therapy
9. Patients with lymphoma that requires immediate cytoreductive therapy
10. Patients on the drugs which are sensitive substrates of CYP2C8 and cannot be discontinued at least one week prior to Cycle 1 Day 1
11. Patients on the drugs which are sensitive substrates of either Poglycoprotein (P-gp) or breast cancer resistance protein (BCRP) and cannot be discontinued at least one week prior to Cycle 1 Day 1
12. Major surgery ≤ 28 days from Cycle 1 Day 1 (major surgery is defined as a procedure requiring general anesthesia)
13. Active infection requiring systemic therapy. Note: Prophylactic use of antibiotics is allowed. Any infection detected during screening period which is resolved adequately according to investigator before the Cycle 1 Day 1, is allowed.
14. Known to be human immunodeficiency virus (HIV) positive or have an acquired immunodeficiency syndrome-related illness
15. Known active or chronic hepatitis B (HbsAg +ve) or hepatitis C infection (HCV antibody +ve)
16. The patient who is expected to require any other form of antineoplastic therapy or targeted therapy while on study.
17. Uncontrolled congestive heart failure (New York Heart Association (NYHA) Class 2-4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, or transient ischemic attack, or pulmonary embolism within 3 months prior to Cycle 1 Day 1
18. Ongoing cardiac dysrhythmias requiring treatment of any grade or treatment of cardiac dysrhythmias in past 3 months, before Cycle 1 Day 1.
19. QTc (Bazzett) interval >460 ms on ECG at screening and/or at Cycle 1 Day 1 pre-dose.
20. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or significant gastritis, active bleeding diatheses, presence of any major medical illness (e.g. renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, or psychiatric illness/social situations or clinically significant laboratory / ECG abnormalities at screening, any or a combination of illnesses, which, in the opinion of the PI, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study
21. Current swab-positive or suspected (under investigation) Covid-19 infection or fever and other signs or symptoms suggestive of Covid-19 infection with recent contact of person(s) with confirmed Covid-19 infection, at screening or Cycle 1 Day 1.
22. History of another primary malignancy within 5 years prior to starting study drug, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ and the disease under study.
23. Positive pregnancy test for women of child-bearing potential (WOCBP) at the screening or enrolment visit
24. Lactating women or WOCBP who are neither surgically sterilized nor willing to use reliable contraceptive methods (hormonal contraceptive, IUD, or any double combination of male or female condom, spermicidal gel, diaphragm, sponge, cervical cap).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
1. First cycle Dose Limiting Toxicities (DLT) | 28 Days
  Assess dose limiliting toxicities of AUR108
Safety of AUR108 as measured by the number of participants with treatment-related adverse events (AE) graded according to NCI CTCAE version 5.0 | Through study completion, an average of 1 year
  Number of participants with TEAEs
Pharmacokinetics Maximum Concentration (Cmax) | Day 1 and Day 17
  Maximum Concentration of AUR108
Pharmacokinetics: Time to Maximum concentration (Tmax) | Day 1 and Day 17
  Tmax in hours
Pharmacokinetics: Area under the curve (AUC) | Day 1 and Day 17
  Area under the curve (AUC) of AUR108 in h* ng/mL
Pharmacokinetics: Terminal elimination half-life | Day 17
  Terminal elimination half-life of AUR 108 in hours
Maximum concentration (Cmax) administered under fasting/fed condition | Day 8
  Compare in fast and fed conditions
Time to Maximum concentration (Tmax) administered under fasting/fed condition | Day 8
  Compare Tmax in fast and fed conditions
Area under curve (AUC) administered under fasting/fed condition | Day 8
  Compare AUC in fast and fed conditions

OTHER OUTCOMES:
PD biomarker assessment | Day 1, Day 2, Day 17 and Day 18
  Change from baseline in biomarker (DHO) levels
Overall Response Rate | Through study completion, an average of 1 year
  Efficacy assessments by Overall Response Rate
Duration of Response | Through study completion, an average of 1 year
  Efficacy assessments by Duration of Response
Progression Free Survival | Through study completion, an average of 1 year
  Efficacy assessments by Progression Free Survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Akhil Kumar, Principal Investigator — Chief Medical Officer
Locations (20):
- India (20):
  - Omega Cancer Hospitals, Visakhapatnam, Andhra Pradesh
  - HCC Happiness Care and Cure Multispeciality Hospital, Ahmedabad, Gujarat
  - Unique Hospital, Surat, Gujarat
  - Kiran Multi Speciality Hospital, Surat, Gujarat
  - Super Specialty Hospital (G.M.C) Srinagar, Srinagar, Jammu and Kashmir
  - KLES Dr Prabhakar Kore Hospital and MRC, Belagavi, Karnataka
  - Amrita Institute of Medical Sciences (AIMS), Kochi, Kerala
  - Sujan Surgical Cancer Hospital and Amravati Cancer Foundation, Amravati, Maharashtra
  - Kolhapur Cancer Centre, Kolhāpur, Maharashtra
  - Mumbai Onco Care Centre, Mumbai, Maharashtra
  - All India Institute of Medical Sciences, Nagpur, Maharashtra
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Center, Pune, Maharashtra
  - MTES Sanjeevan Hospital, Pune, Maharashtra
  - All India Institute of Medical Sciences, Delhi, New Delhi
  - Sparsh Hospital and Critical Care (P) Ltd., Bhubaneswar, Odisha
  - MNJ Institute of Oncology and Regional Cancer Centre, Hyderabad, Telangana
  - Tata Medical Center, Kolkata, West Bengal
  - Post Graduate Institute of Medical Education & Research,, Chandigarh
  - Rajiv Gandhi Cancer Institute and Research Centre, Delhi

IPD SHARING:
Plan to Share IPD: No